CLINICAL TRIAL: NCT00247559
Title: A Phase II, Multi-Centre, Randomised, Double-blind, Dose-Ranging Study Comparing the Efficacy and Safety of a Single Treatment With 15, 30 or 45 Units (Per Eye) of Dysport to Placebo in the Symptomatic Treatment of Lateral Canthal Lines (Crow's Feet)
Brief Title: Botulinum Type A Toxin in the Treatment of Lateral Canthal Lines (Crow's Feet)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-97-52120-723; 2004-001421-17 (EudraCT Number)
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Lateral Canthal Lines
Keywords: crow's feet; cosmesis; ageing
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
Despite the wealth of information in the literature regarding the cosmetic applications of botulinum type A toxin (BoNT-A), and the widespread use of the BoNT-A for cosmetic applications, the number of randomised, controlled clinical trials is small. Much of the published information is based on open-label studies or anecdotal data. Of the robust trial data that is available, the vast majority relates to the treatment of glabellar lines, and there is little data available regarding the use of BoNT-A in lateral canthal lines. This study aims to determine the optimum dose for the use of BoNT-A in this area.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 to 65 years of age.
* In the opinion of the Investigator moderate to severe lateral canthal lines (crow's feet) during maximum smile on both sides of the face.
* In the opinion of the Investigator mild to severe lateral canthal lines (crow's feet) at rest on both sides of the face.

Exclusion Criteria:

* Any prior surgery affecting the orbicularis oculi muscle, prior blepharoplasty or brow lift, or any prior cosmetic procedures or scars that may interfere with the evaluation of the study results.
* Previous insertion of any non-absorbable material in the periorbital region or facial treatment with augmentation material within 12 months prior to screening.
* Any prior treatment with botulinum toxin (of any serotype).
* Previous treatment with lasers for skin resurfacing or treatment with deep chemical peels within 12 months prior to screening.
* Inability to substantially lessen the lateral canthal lines by physically spreading them apart.
* Facial conditions that could affect safety or efficacy results such as: active infection or other skin problem in the periorbital area (e.g. acute acne lesions or ulcers); history of facial nerve palsy; marked facial asymmetry; ptosis; excessive dermatochalasis; deep dermal scarring; thick sebaceous skin; photodamage etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2004-05; Primary Completion 2005-04-08 (Actual); Study Completion 2005-04-08 (Actual)

PRIMARY OUTCOMES:
Change in severity of crow's feet at maximum smile at week 4, compared to baseline, assessed photographically by independent panel

SECONDARY OUTCOMES:
At week 2,4,8,12,16,20,24, compared to baseline: change in severity of crow's feet at rest & max. smile, assessed by investigator & independent panel (photographically); change in patient satisfaction with appearance of crow's feet & general appearance

CONTACTS AND LOCATIONS:
Overall Officials: UK Medical Director, Study Director — Ipsen
Locations (9):
- France (3):
  - Clinique Bel Air, Bordeaux
  - Centre Hospitalier Universitaire de Nice, Nice
  - Service de Chirurgie Maxillo Faciale, Saint-Cloud
- Germany (3):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Dermatologie, Stadt. Klinikum Dresden-Friedrichstadt, Dresden
  - Universitats - Hautklinik, Homburg
- United Kingdom (3):
  - The Cambridge Private Hospital, Cambridge, England
  - Harley Street, London, England
  - The Golden Jubilee National Hospital, Clydebank, Scotland